CLINICAL TRIAL: NCT05660603
Title: Circum-Psoas Blocks Versus Combined Lumbar and Sacral Plexus Blocks for Sensory Level and Postoperative Analgesia Obtained in Hip Fracture Surgery
Brief Title: Circum-Psoas Blocks Versus Combined Lumbar and Sacral Plexus Blocks in Hip Fracture Surgery
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Zagazig University (Other Government)
Responsible Party: Principal Investigator, Shereen Elsayed Abd Ellatif, associate professor of anesthesia and surgical intensive care, Zagazig University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 10177/13/12/2022
Record Dates: First submitted 2022-12-13; First posted 2022-12-21 (Actual); Last update posted 2025-07-17 (Actual); Status verified 2025-07

CONDITIONS: Hip Fractures
Keywords: circum-psoas blocks; lumbar plexus block; sacral plexus block; hip fracture surgery
MeSH Terms: conditions — Hip Fractures | interventions — Ultrasonography

STUDY DESIGN:
Intervention Model Description: The patients will be divided randomly by a computer-generated randomization table into three groups :
  Group C :(Control group) patients will receive standard general anesthesia. Group LSP: patients will receive standard general anesthesia followed by combined lumbar and sacral plexus blocks with 40 ml of bupivacaine 0.25%.
  Group CP: patients will receive standard general anesthesia followed by circum-psoas block with 40 ml of bupivacaine 0.25%.
Who Masked: Participant, Outcomes Assessor
Masking Description: double-blinded(participants and outcome assessors)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- control group (Placebo Comparator): patients will be operated on under general anesthesia
  Interventions: Other: control
- LSP group (lumbar and sacral plexus block) (Active Comparator): patients will receive ultrasound-guided combined lumbar and sacral plexus blocks with 40 ml of 0.25% of bupivacaine.
  Interventions: Procedure: LSP; Device: Ultrasound
- CP group (circum-psoas block) (Active Comparator): patients will receive ultrasound-guided circum-psoas blocks with 40 ml of 0.25% of bupivacaine.
  Interventions: Procedure: CP; Device: Ultrasound

INTERVENTIONS:
Other: control — patients will receive standard general anesthesia
  Arms: control group
Procedure: LSP — patients will receive standard general anesthesia followed by ultrasound-guided combined lumbar and sacral plexus blocks with 40 ml of bupivacaine 0.25%.
  Arms: LSP group (lumbar and sacral plexus block)
Procedure: CP — patients will receive standard general anesthesia followed by ultrasound-guided circum-psoas blocks with 40 ml of bupivacaine 0.25%.
  Arms: CP group (circum-psoas block)
Device: Ultrasound — ultrasound
  Arms: CP group (circum-psoas block); LSP group (lumbar and sacral plexus block)

SUMMARY:
Hip fracture (HF) is one of the major worldwide problems that constitute a significant mortality rate, ranging from 14- 36% in the first year after injury, and is associated with profound temporary and sometimes permanent impairment of independence and quality of life in the geriatric population. Surgical treatment is considered the best option for patients with hip fractures,s especially in the elderly, however, it is associated with moderate to severe postoperative pain.

Pain is one of the main factors limiting ambulation, increasing the risk of thromboembolism by immobility and causing metabolic changes that affect other systems. Therefore, individualized pain management with the use of appropriate analgesic techniques is of paramount importance. Moreover, early intervention of rehabilitation aiming at a better postoperative recovery may reduce the length of hospital stay and return to daily. Effective pain management is one of the crucial components in enhanced recovery after surgery (ERAS).

• Numerous regional anesthetic techniques have been used to provide analgesia following hip fracture surgery, including intrathecal morphine, epidural analgesia, fascia iliaca block, lumber plexus block, and sacral plexus block, however, each of these techniques has specific limitations that prevent them from being the analgesic technique of choice for hip fracture surgery.

To our knowledge, there is no study done to compare circum-psoas block versus the combined lumbar and sacral plexus blocks as pre-emptive analgesia in patients undergoing hip fracture surgery under general anesthesia.

DETAILED DESCRIPTION:
The acetabulum and the head of the femur combine to produce a traditional ball and socket joint in the hip. Both the lumbar (L1-L4) and sacral (L4-S4) plexuses innervate the hip joint, and its sensory innervation is from the femoral (FN), obturator, and sciatic nerves with contribution from superior gluteal nerve and nerve to quadratus femoris. Cutaneous innervation is by lateral femoral cutaneous (LFCN), subcostal iliohypogastric nerve, and the superior cluneal nerves which predominately arise from the dorsal rami of L1.

Hip fracture is a major worldwide public health problem in elderly patients aged 65 years and over with an incidence of more than 1.6 million worldwide each year. Furthermore, the total number is expected to exceed 6 million by 2050. Generally, early surgical repair within 48-72 hours after admission is recommended according to the treatment guideline, however, elderly patients with hip fractures commonly have several comorbidities, which make these patients more liable to a high risk of morbidity and mortality after surgery. Pain, both before and during the first 24 hours of surgery is usually reported as severe by most patients therefore, one of the keys to a patient's recovery following hip fracture surgery, is effective postoperative pain management. Recently, the concept of pain relief with multimodal analgesia and regional anesthesia plays a vital role in postoperative analgesia minimizing opioid consumption and reducing the time to early mobilization. The acetabulum and the head of the femur combine to produce a traditional ball and socket joint in the hip. The lumbar (L1-L4) and sacral (L4-S4) plexuses both innervate the hip joint, and its sensory innervation is from the femoral (FN), obturator, and sciatic nerves with contribution from superior gluteal nerve and nerve to quadratus femoris. Cutaneous innervation is by lateral femoral cutaneous (LFCN), subcostal iliohypogastric nerve, and the superior cluneal nerves which predominately arise from the dorsal rami of L1.

Hip fracture is a major worldwide public health problem in elderly patients aged 65 years and over with an incidence of more than 1.6 million worldwide each year. Furthermore, the total number is expected to exceed 6 million by 2050. Generally, early surgical repair within 48-72 hours after admission is recommended according to the treatment guideline, however, elderly patients with hip fractures commonly have several comorbidities, which make these patients more liable to a high risk of morbidity and mortality after surgery. Pain, both before and during the first 24 hours of surgery is usually reported as severe by most patients therefore, one of the keys to a patient's recovery following hip fracture surgery, is effective postoperative pain management. Recently, the concept of pain relief with multimodal analgesia and regional anesthesia plays a vital role in postoperative analgesia minimizing opioid consumption and reducing the time to early mobilization. Several regional anesthetic techniques have been recommended, including intrathecal morphine, patient-controlled epidural analgesia, and various peripheral nerve blocks techniques; however, to obtain complete sensory loss for hip fracture surgery, it's required to block the branches of both lumbar and sacral plexuses, although there remains no single technique that reliably acquires this. Moreover, each of these techniques has specific limitations that prevent them from being the analgesic technique of choice for hip fracture surgery.

The ultrasound-guided lumbar plexus block results in the blockade of the FN, LFCN, and obturator nerve while the sacral plexus block results in the blockade of the sciatic nerve, superior and inferior gluteal nerves, posterior cutaneous nerve of the thigh, and the inferior hypogastric plexus. Thus, the combination of lumbar plexus and sacral plexus blocks results in complete analgesia of the ipsilateral lower limb in the perioperative period.

Circum-psoas blocks is a new sonar-guided fascial block technique proposed by Huili et al., where the two main branches of the lumbar plexus (FN and LFCN) can be blocked by local anesthetic (LA) injection posterior to transversalis fascia (TF) and around the anterolateral edge of psoas muscle (PM) just cranial to iliac crest. Furthermore, cranial spread along TF may lead to a lower thoracic paravertebral block through the medial arcuate ligament. On the other hand, the obturator nerve and lumbosacral trunk could be blocked if the LA is injected at the level of L5/S1 into the retro-psoas space and around the posterior edge of PM.

Our study will be designed to evaluate and compare the impact of combined lumbar and sacral plexus blocks and circum-psoas blocks for sensory level and achievement of postoperative analgesia for patients undergoing hip fracture surgery under general anesthesia.

ELIGIBILITY:
Inclusion Criteria:

* Patient acceptance.
* BMI ≤ 30 kg/m2
* ASA I-III.
* First unilateral surgery for hip fracture including femoral neck, intertrochanteric or subtrochanteric fracture.
* Patient with planned hip fracture surgery within 24-72 hours under general anesthesia.

Exclusion Criteria:

* Multiple trauma, multiple fractures, or pathological fractures
* Prosthetic fracture or usage of bone-cement fixation in the surgery.
* Scheduled for bilateral hip fracture surgery.
* Pre-existing neurological deficit in the lower extremity
* Contraindication for peripheral nerve block (infection at the site of needle insertion, coagulopathy, allergy to local anesthetics used)
* History of chronic pain and taking analgesics
* History of cognitive dysfunction or mental illness

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 63 (Estimated)
Dates: Start 2022-12-20 (Actual); Primary Completion 2026-02-01 (Estimated); Study Completion 2026-04-01 (Estimated)

PRIMARY OUTCOMES:
Assess change of Visual analogue scale (VAS) | at 30 minutes, 2 hours, 4, 6,12, 24 hours postoperatively
  On a scale of 0-10, the patient will learn to quantify postoperative pain where 0= No pain and 10= Maximum worst pain

SECONDARY OUTCOMES:
Assess sensory block levels | at 2 hours postoperatively
  by using alteration of pinprick sensation compared to the contralateral side on the dermatomes supplied by blocked nerves
Total dose of rescue analgesia | in the first 24 hour postoperatively
  once the VAS score will be ≥ 3, rescue analgesia in the form of 1 μg/kg fentanyl will be given and the total dose consumed will be recorded

CONTACTS AND LOCATIONS:
Locations (1):
- Shereen E Abd Ellatif, Zagazig, Alsharqia, Egypt

IPD SHARING:
Plan to Share IPD: Yes
planned after the completion of the study and publication
Supporting Information: Study Protocol, SAP, CSR
Time Frame: planned after the completion of the study and publication
Access Criteria: contact with principal investigator

REFERENCES:
- [Background] Roche JJ, Wenn RT, Sahota O, Moran CG. Effect of comorbidities and postoperative complications on mortality after hip fracture in elderly people: prospective observational cohort study. BMJ. 2005 Dec 10;331(7529):1374. doi: 10.1136/bmj.38643.663843.55. Epub 2005 Nov 18. PMID 16299013
- [Background] Bendtsen TF, Pedersen EM, Haroutounian S, Soballe K, Moriggl B, Nikolajsen L, Hasselstrom JB, Fisker AK, Strid JM, Iversen B, Borglum J. The suprasacral parallel shift vs lumbar plexus blockade with ultrasound guidance in healthy volunteers--a randomised controlled trial. Anaesthesia. 2014 Nov;69(11):1227-40. doi: 10.1111/anae.12753. Epub 2014 Jun 28. PMID 24974961
- [Background] Petchara S, Paphon S, Vanlapa A, Boontikar P, Disya K. Combined Lumbar-Sacral Plexus Block in High Surgical Risk Geriatric Patients undergoing Early Hip Fracture Surgery. Malays Orthop J. 2015 Nov;9(3):28-34. doi: 10.5704/MOJ.1511.004. PMID 28611906
- [Background] Li H, Shi R, Shao P, Wang Y. Evaluation of Sensory Loss Obtained by Circum-Psoas Blocks in Patients Undergoing Total Hip Replacement: A Descriptive Pilot Study. J Pain Res. 2022 Mar 29;15:827-835. doi: 10.2147/JPR.S354829. eCollection 2022. PMID 35378731